CLINICAL TRIAL: NCT05950659
Title: Prevention of Foot Ulcer Recurrence in Individuals Who Are at High-risk for Diabetic Foot Complications Using the Orpyx Sensory Insole System: a Multisite, Randomized, Controlled Trial
Brief Title: WIREDUP: Wearable Insoles for Recurrent Diabetic Ulcer Prevention
Acronym: WIREDUP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orpyx Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WIREDUP
Record Dates: First submitted 2023-07-11; First posted 2023-07-18 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Diabetes; Peripheral Neuropathy; Diabetic Foot; Diabetic Foot Ulcer
Keywords: Remote Patient Monitoring; Sensor-based Monitoring; Sensory Insoles
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Nervous System Diseases; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental)
  Interventions: Device: Orpyx Sensory Insole System
- Control (No Intervention)

INTERVENTIONS:
Device: Orpyx Sensory Insole System — The Orpyx Sensory Insoles System uses Orpyx Sensory Technology: a powered limb overload warning technology intended for monitoring physiologic parameters, such as plantar pressure, temperature, motion, and adherence, and providing real-time cues for pressure offloading
  Arms: Intervention

SUMMARY:
The primary aim of this study is to demonstrate the impact of the Orpyx® Sensory Insoles (Orpyx Medical Technologies Inc., Calgary AB, Canada) ("Orpyx" or "the Company") as an adjunct to the standard of care (SOC), as compared to SOC alone, on reducing plantar ulceration incidence in individuals who are at risk for developing diabetic foot complications.

The secondary aims of this study are to evaluate participant quality of life, participant engagement, and economic impact, including cost-effectiveness and cost-utility. The study will also use the unique data set collected (plantar pressure, temperature, step count, movement and adherence feedback) to identify foot-loading histories that either lead to or prevent the development of ulceration in the diabetic foot.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Type 1 or 2 diabetes
* Clinically diagnosed neuropathy via Neuropathy Monofilament Test
* Qualification as a "high-risk participant," meaning a recent history (<12 months) of a healed diabetic neuropathic ulceration on the weight-bearing surface of one or both feet (this includes the plantar distal toe surface)
* Complete healing of any previous foot ulcers, as defined by complete re-epithelialization of that ulcer which is confirmed by two medical exams that occur at least two weeks apart (V0 and V1)
* Ability to walk independently (without use of wheelchair) for 30 steps. Use of a walker or cane is acceptable as long as the participant can walk for at least 30 steps.
* Aged >18 years
* Ability to understand all study requirements and have a life expectancy greater than the study duration
* Vascular assessment (i.e., ABI, segmental pressure) that demonstrates the participant has adequate lower extremity perfusion
* Subject is willing and able to maintain the required offloading (as applicable for the location of the healed ulcer)
* Subject is willing and able to wear the Orpyx Sensory Insoles during ambulatory activity and at home during waking hours, and for a minimum of 5 hours per day
* Compatibility of the device with the participant's footwear
* Most recent HbA1c level of < 12.0% (in the last 12 months)
* Amputations, if present, are compatible with the use of insoles

Exclusion Criteria:

* Active ulcer or presence of other open chronic wound (on foot or other body surface), regardless of etiology (e.g., vasculitis, neoplasms, or hematological disorders)
* History of known non-neuropathic foot ulcer (e.g., arterial, or venous insufficiency ulcer)
* Presence of severe vascular disease (refer to acceptable ABI parameters in inclusion criteria)
* Dementia
* Psychiatric illness or social situations that would limit compliance with the study
* Serious underlying balance dysfunction, regardless of etiology
* Significant cardiopulmonary or other systemic disease limiting the participant's ability to walk at least 30 steps or to stand for an amount of time equal to or greater than five (5) minutes
* Current participation in another clinical investigation of a medical device or a drug; or participation in such a study within 30 days prior to study enrolment
* Osteomyelitis or gangrene of the lower extremity
* Uncorrected plantar Charcot neuroarthropathy
* Bunion which would predispose ulcer formation (clinician discretion)
* Extreme equinus
* Hallux valgus
* Hallux rigidus / limitus
* HbA1c levels >= 12%
* At the start of V1, and prior to randomization, the subject no longer meets the entrance criteria (inclusion and exclusion)
* Any condition that would affect or limit the ability to properly fit both shoes with the device under study
* Subject has a history of intercurrent illness or conditions that would compromise the safety of the subject or their ability to participate in the study
* Amputations on the foot which the clinician deems incompatible with the insoles (i.e., those that require additive insole modifications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Plantar ulcer recurrence | 12 months

IPD SHARING:
Plan to Share IPD: No